CLINICAL TRIAL: NCT02504515
Title: Evaluating Treatment With Homeopathy, Acupuncture, and Anthroposophic Medicine in Improving the Quality of Life for Women Treated at the Public Unified Healthcare System
Brief Title: Effect of Homeopathy, Acupuncture or Anthroposophic Medicine in Women's Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Rubens Lene Carvalho Tavares, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22858113.9.0000.5149
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Anxiety; Depression; Premenstrual Tension; Hot Flashes; Muscular Diseases
MeSH Terms: conditions — Anxiety Disorders; Depression; Premenstrual Syndrome; Hot Flashes; Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Homeopathy (Active Comparator)
  Interventions: Other: World Health Organization Quality of Life Bref Questionnaire
- Allopathy homeopathy control (Active Comparator)
  Interventions: Other: World Health Organization Quality of Life Bref Questionnaire
- Acupuncture (Active Comparator)
  Interventions: Other: World Health Organization Quality of Life Bref Questionnaire
- Allopathy acupuncture control (Active Comparator)
  Interventions: Other: World Health Organization Quality of Life Bref Questionnaire
- Anthroposophic medicine (Active Comparator)
  Interventions: Other: World Health Organization Quality of Life Bref Questionnaire
- Allopathy anthroposophy control (Active Comparator)
  Interventions: Other: World Health Organization Quality of Life Bref Questionnaire

INTERVENTIONS:
Other: World Health Organization Quality of Life Bref Questionnaire — The World Health Organization Bref (WHOQOL-BREF) questionnaire will be applied in three different moments: Baseline, after 6 months, and after 12 months.
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.

SUMMARY:
Patients will be randomly assigned to two separate groups. Both patient groups will be evaluated using the WHOQOL-BREF questionaire. Evaluations will be carried out just before the study begins and at intervals of six months during a period of one year for a total of three evaluations. Group one will be made up of patients who will begin homeopathy or acupuncture or anthroposophic medicine treatment and patients from group two will start homeopathy or acupuncture or anthroposophic medicine six months after the beginning of the study. Each one of these three research branches will be done independently (Homeopathy versus control; Acupuncture versus control; Anthroposophic Medicine versus control). Conventional medical treatment will be available for all patients in both groups. A data sheet will be filled out on each patient with data as to age, education level, marital status and the patient's own perception of their health status. During the interviews the interviewer will have no influence whatsoever over the respondents' answers. Integrative/complementary or traditional medicine doctors do not participate in the research and will not be informed about which patients are participating in this project, and as such the research will be blinded for these doctors. Minitab software, version 16, was used for sample calculation through the module Power and Sample Size. Sample calculation option for paired t-tests before and after intervention demonstrated the need to randomize 906 patients: 450 patients for homeopathy branch (225 patients in the homeopathy group and 225 patients in the control group), 228 patients for acupuncture branch (114 patients in the acupuncture group and 114 patients in the control group), and 228 patients for anthroposophic medicine branch (114 patients in the anthroposophic medicine group and 114 patients in the control group).

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Patients with chronic diseases

Exclusion Criteria:

* Women below 18 years of age
* Previous treatment with homeopathy (for homeopathy versus control branch)
* Previous treatment with acupuncture (for acupuncture versus control branch)
* Previous treatment with anthroposophic medicine (for anthroposophic medicine versus control branch)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | one year

SECONDARY OUTCOMES:
Quality of life | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil